CLINICAL TRIAL: NCT05566080
Title: Preoperative Identification of the Histologically "Vulnerable" Plaque Using Non-invasive Imaging, Biomechanical Assessment and Baroreflex Evaluation in Patients With Severe Carotid Stenosis
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Pavia (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: GR-2018-12366862
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Carotid Artery Plaque; Diagnosis
Keywords: carotid stenosis; ultrasonic imaging; finite element analysis
MeSH Terms: conditions — Carotid Stenosis; Disease | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — carotid atherosclerotic plaque
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Carotid endarterectomy — Patients who have a significant carotid stenosis and who undergo surgical carotid endarterectomy

SUMMARY:
Carotid artery stenosis due to atherosclerotic plaques accounts for an important cause of ischemic stroke. Current research seeks to risk stratify asymptomatic patients by characterizing rupture-prone plaques. Currently no single imaging modality can reliably identify those plaques before surgery. Recently, the 3D ultrasound (US) and the assessment of the mechanical stress on the vessel wall have been proposed as non-invasive tools that could play a role in the diagnostic work-up. Data of histological validation, however, are still needed. In this research, 3D US, non-invasive elastography, Finite Element Analysis of computed tomography angiography images and the study of the autonomic cardiovascular control will be used to identify preoperatively the vulnerable plaque in patients undergoing carotid endarterectomy. The results will be compared to that of histology of the removed plaque, aiming to provide a validation to each method for a possible application in the daily practice.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years;
* signed informed consent.

Exclusion Criteria:

* medical conditions limiting expected survival to <1 year;
* patients with significant uncontrolled or unstable medical condition (heart failure or angina pectoris class NYHA III-IV, cardiac surgery in the previous 30 days, left ventricular ejection fraction <30%, severe chronic obstructive pulmonary disease, myocardial infarction in the previous 30 days, coronary heart disease with revascularization indication, that is, the common trunk or more than two coronary vessels);
* tracheostomy;
* paralysis of the laryngeal nerve contralateral to the carotid stenosis;
* women of childbearing potential;
* inability to give informed consent;
* patients presenting contraindications to perform a CTA examination of neck vessels with contrast medium;
* patients with medical history of stroke/TIA within the previous 6 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CEA for a 70-99% asymptomatic stenosis according to ECST measurement of the internal carotid artery at Unit of Vascular Surgery, IRCCS Policlinico San Donato.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Plaque vulnerability | Through study completion, an average of 3 years
  To assess the correlation between the result of 3D US in identifying preoperatively the features of vulnerable plaque (plaque volume; presence of a lipidic core/intraplaque hemorrhage/plaque ulceration; fibrous cap thickness) and that of the histological analysis, in patients who will undergo CEA for a 70-99% carotid stenosis. To assess the correlation between the US-SE parameters to plaque vulnerability, as defined by the histological analysis.
Plaque vulnerability | Through study completion, an average of 3 years
  To assess the state of the autonomic function and cardiovascular control in patients undergoing CEA and check if there is a relation with the histological analysis of the carotid plaque after CEA.
Plaque vulnerability | Through study completion, an average of 3 years
  To develop software routines to process US B-mode and US-SE images; to determine the mechanical stress patterns on the vessel wall by the different types of carotid plaques through the FEA of preoperative CTA scans of the recruited patients, and their correlation with the plaque histology and 3D US images. relation with the histological analysis of the carotid plaque after CEA.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kolos I, Troitskiy A, Balakhonova T, Shariya M, Skrypnik D, Tvorogova T, Deev A, Boytsov S; Aggressive Medical Treatment Evaluation for Asymptomatic Carotid Artery Stenosis (AMTEC) Study Group. Modern medical treatment with or without carotid endarterectomy for severe asymptomatic carotid atherosclerosis. J Vasc Surg. 2015 Oct;62(4):914-22. doi: 10.1016/j.jvs.2015.05.005. PMID 26410046
- [Background] Spence JD. Endarterectomy vs. stenting vs. medical therapy. Int J Stroke. 2016 Jul;11(5):500-1. doi: 10.1177/1747493016643552. Epub 2016 Apr 11. PMID 27256474
- [Background] Gupta A, Baradaran H, Schweitzer AD, Kamel H, Pandya A, Delgado D, Dunning A, Mushlin AI, Sanelli PC. Carotid plaque MRI and stroke risk: a systematic review and meta-analysis. Stroke. 2013 Nov;44(11):3071-7. doi: 10.1161/STROKEAHA.113.002551. Epub 2013 Aug 29. PMID 23988640
- [Background] Huibers A, de Borst GJ, Wan S, Kennedy F, Giannopoulos A, Moll FL, Richards T. Non-invasive Carotid Artery Imaging to Identify the Vulnerable Plaque: Current Status and Future Goals. Eur J Vasc Endovasc Surg. 2015 Nov;50(5):563-72. doi: 10.1016/j.ejvs.2015.06.113. Epub 2015 Aug 19. PMID 26298222
- [Background] AlMuhanna K, Hossain MM, Zhao L, Fischell J, Kowalewski G, Dux M, Sikdar S, Lal BK. Carotid plaque morphometric assessment with three-dimensional ultrasound imaging. J Vasc Surg. 2015 Mar;61(3):690-7. doi: 10.1016/j.jvs.2014.10.003. Epub 2014 Dec 9. PMID 25499716
- [Background] Mahmood B, Ewertsen C, Carlsen J, Nielsen MB. Ultrasound Vascular Elastography as a Tool for Assessing Atherosclerotic Plaques - A Systematic Literature Review. Ultrasound Int Open. 2016 Nov;2(4):E106-E112. doi: 10.1055/s-0042-115564. Epub 2016 Oct 13. PMID 27896334
- [Background] Tsekouras NS, Katsargyris A, Skrapari I, Bastounis EE, Georgopoulos S, Klonaris C, Bakoyiannis C, Bastounis EA. The role of carotid plaque echogenicity in baroreflex sensitivity. J Vasc Surg. 2011 Jul;54(1):93-9. doi: 10.1016/j.jvs.2010.11.121. Epub 2011 Mar 31. PMID 21458208
- [Background] Ricotta JJ, Aburahma A, Ascher E, Eskandari M, Faries P, Lal BK; Society for Vascular Surgery. Updated Society for Vascular Surgery guidelines for management of extracranial carotid disease. J Vasc Surg. 2011 Sep;54(3):e1-31. doi: 10.1016/j.jvs.2011.07.031. PMID 21889701
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Pagani M, Montano N, Porta A, Malliani A, Abboud FM, Birkett C, Somers VK. Relationship between spectral components of cardiovascular variabilities and direct measures of muscle sympathetic nerve activity in humans. Circulation. 1997 Mar 18;95(6):1441-8. doi: 10.1161/01.cir.95.6.1441. PMID 9118511
- [Background] van Engelen A, Wannarong T, Parraga G, Niessen WJ, Fenster A, Spence JD, de Bruijne M. Three-dimensional carotid ultrasound plaque texture predicts vascular events. Stroke. 2014 Sep;45(9):2695-701. doi: 10.1161/STROKEAHA.114.005752. Epub 2014 Jul 17. PMID 25034714
- [Background] Sadat U, Li ZY, Young VE, Graves MJ, Boyle JR, Warburton EA, Varty K, O'Brien E, Gillard JH. Finite element analysis of vulnerable atherosclerotic plaques: a comparison of mechanical stresses within carotid plaques of acute and recently symptomatic patients with carotid artery disease. J Neurol Neurosurg Psychiatry. 2010 Mar;81(3):286-9. doi: 10.1136/jnnp.2009.190363. Epub 2009 Nov 25. PMID 19939857
- [Background] Simel DL, Samsa GP, Matchar DB. Likelihood ratios with confidence: sample size estimation for diagnostic test studies. J Clin Epidemiol. 1991;44(8):763-70. doi: 10.1016/0895-4356(91)90128-v. PMID 1941027